CLINICAL TRIAL: NCT01160939
Title: Assessment and Monitoring of Patients in Medium-term Heart Transplant Candidates Undergoing Low-intensity Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: DYYUNIFESP
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2009-11

CONDITIONS: Heart Failure
Keywords: Exercise; heart failure; rehabilitation
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: low intensity exercise — exercise protocol with six stages of exercise (1. upper limbs, 2. inferiors, 3. walk 35 m, 4. ½ flight of stairs, 5. walk 200 m 6. a flight of stairs) with intensity between 2-6 metabolic equivalents

SUMMARY:
Objectives: To study the behavior and cardiovascular safety protocol to the front low-intensity exercise in patients with heart failure (HF) severe, awaiting heart transplantation. Methods: The investigators studied 21 patients with severe HF on the list for a heart transplant at the University Hospital of UNIFESP. After evaluation, patients underwent exercise protocol with six stages of exercise (1. upper limbs, 2. inferiors, 3. walk 35 m, 4. ½ flight of stairs, 5. walk 200 m 6. a flight of stairs) with intensity between 2-6 metabolic equivalents. These also were followed for an average period of 17 months as the clinical complications and death. Results: From the patients studied, three were not able to perform the full protocol, and the variables body mass index, maximal inspiratory and expiratory pressure measurement (Pimáx and Pemáx, cmH2O) and number of previous admissions, showed the most divergent behavior of the sample studied. A greater increase in heart rate, double product and scale of perceived exertion during step 5 was observed during the protocol. Blood pressure levels showed little change between stages, and there was no arrhythmias incidence increase (kappa = 0.552) compared to effort. A positive correlation scale was perceived in exertion walking distance of 200m, with systolic blood pressure (r = 0.4, p = 0.02). Overall observed lower values of maximal inspiratory pressure and increased blood pressure and elevated heart rate in patients with death outcome. Conclusion: Cardiovascular behavior against exercise protocol was well tolerated and safe, but suggests need for monitoring. Information collected at initial clinical evaluation associated with decompensation and death, and may help stratify these patients.

ELIGIBILITY:
Inclusion Criteria:

* heart failure severe, awaiting heart transplantation

Exclusion Criteria:

* decompensated heart failure
* vasoactive drugs
* unstable angina
* severe stenosis or insufficiency valvular
* recent surgery
* morbid obesity

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-11; Primary Completion 2006-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil